CLINICAL TRIAL: NCT02332304
Title: Amniotic Fluid Optical Density Determination Between 28 and 36 6/7 Weeks of Pregnancy and Its Relationship With the Diagnosis of Neonatal Respiratory Distress Syndrome.
Brief Title: Amniotic Fluid Optical Density Determination as a Test for Assessment of Fetal Lung Maturity.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research, Saint Thomas Hospital, Panama
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MHST2014-02
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preterm fetus (Other): Patients with pregnancies between 26 and 36 6/7 weeks of pregnancy. Before the birth, a sample of amniotic fluid was taken and analyzed using optical density at 650nm. A value above 0.15 was considered an indication of fetal lung maturity.
  Interventions: Procedure: Preterm fetus

INTERVENTIONS:
Procedure: Preterm fetus — A sample of amniotic fluid was taken before the birth of fetus between 26 and 36 6/7 weeks of pregnancy.

SUMMARY:
To determine the relationship between the result of amniotic fluid optical density between 26 and 36 6/7 weeks of pregnancy and the risk of developing neonatal respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between 26 and 36 6/7 weeks.

Exclusion Criteria:

* Problems in the handling of the amniotic fluid sample that prevented the calculation of the optical density.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Respiratory Distress Syndrome, Newborn | 1 month
  Diagnosis of Respiratory Distress Syndrome in the neonatal period. The diagnosis was made by the neonatologist in charge (using clinical and radiological parameters).

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Study Director — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Panama